CLINICAL TRIAL: NCT06583408
Title: The REgistry of Very Early Estrogen and AnovuLation
Acronym: REVEAL
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Chrisandra L. Shufelt, MD, Chair and Professor of Medicine, Mayo Clinic
Other Study IDs: 24-000952
Record Dates: First submitted 2024-08-22; First posted 2024-09-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Hypothalamic Amenorrhea, Functional; Hypothalamic Amenorrhea; Functional Hypogonadotropic Hypogonadism
Keywords: Anovulation; Estrogen Loss; Hypoestrogenemia
MeSH Terms: conditions — Anovulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with > 3 months amenorrhea: Women aged 18-40 years old with a diagnosis of functional hypothalamic amenorrhea, or lab results that are within the inclusion criteria.
  Interventions: Other: Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24); Other: REVEAL Questionnaire

INTERVENTIONS:
Other: Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) — Subjects will complete the ASA food diary for 2 weekdays and 1 weekend day
Other: REVEAL Questionnaire — Subjects will complete the REVEAL questionnaire form. This form includes questions about current and past medical history, including reproductive history, lifestyle specifics, and assessment of current health status.

SUMMARY:
The purpose of this study is to to build a registry of women with early estrogen loss due to Functional Hypothalamic Amenorrhea (FHA) to understand the prevalence, racial and ethnic diversity of this condition.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more months of consecutive amenorrhea with a diagnosis of functional hypothalamic amenorrhea or screening hormones consistent with functional hypothalamic amenorrhea including but not limited to:

  * Estradiol: < 50pg/mL
  * LH: < 10 IU/mL
  * FSH: < 10 IU
  * Testosterone: 2 - 45 ng/dL
  * Free Testosterone: 0.1 - 6.4 pg/mL
  * FT4: 0.93 - 1.70 ng/dL
  * Prolactin: < 20 ng/mL
  * AMH: > 1 ng/mL
  * Urine or serum human chorionic gonadotropin: Negative
* LH:FSH Ratio <1
* No signs of male-like hair growth on the upper lip, chin, chest, abdomen, buttocks, or back
* Does not have a diagnosis for secondary amenorrhea, including prolactinoma, PCOS, premature ovarian insufficiency, pituitary surgery, infection, or infarction
* Premenopausal status determined by WISE criteria
* Able to give informed consent
* Able to read English

Exclusion Criteria:

* Parturition/lactating in the last 6-12 months
* Lack of consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study subjects are women aged 18-40 years old with a diagnosis of Functional Hypothalamic Amenorrhea (FHA) or lab results that are within the inclusion criteria. To ensure accurate case ascertainment before enrollment into the study, volunteers must have a diagnosis of FHA from a provider with previously performed lab tests, which will be reviewed and adjudicated by a women's health expert to confirm a diagnosis of FHA. If the potential participant doesn't have access or cannot obtain the required lab results, they can contact the study team to receive an at-home finger-stick hormone test (U.S. Specialty Labs) paid for by the study.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Study Participants | 5 years
  Establish and maintain a comprehensive registry of patients diagnosed with Functional Hypothalamic Amenorrhea (FHA). This registry will include detailed demographic information, clinical data, and longitudinal follow-up to track the prevalence, underlying causes, risk factors, and prognosis of FHA. It will also facilitate the collection of data on racial and ethnic disparities, lifestyle factors, psychological stressors, hormonal imbalances, and the impact of various treatment interventions on long-term health outcomes collected through questionnaires done at baseline and yearly.

SECONDARY OUTCOMES:
Assessing the Impact of Amenorrhea on Women's Health: Symptoms, Care Experiences, and Work Productivity | 5 years
  Improve understanding of women's overall experience of Functional Hypothalamic Amenorrhea (FHA) by documenting the types of care received, frequency and quality of healthcare interactions, and patient satisfaction with the care provided. This includes detailed assessments of specific treatments or therapies received, the involvement of multidisciplinary care approaches, and the extent of follow-up care. Additionally, to quantify the impact of FHA on lost work productivity, including the number of workdays missed, impact on work performance, and economic burden associated with amenorrhea-related issues, measured at baseline and then yearly using questionnaires.
Impact of Social, Early Life, and Pregnancy Factors on Functional Hypothalamic Amenorrhea | 5 years
  Enhance the understanding of how social determinants of health-such as socioeconomic status, education, access to healthcare, and community environment-contribute to the development of Functional Hypothalamic Amenorrhea (FHA). Additionally, the study will explore the impact of childhood adversity, including exposure to trauma, abuse, neglect, or chronic stress, on the likelihood of developing FHA. The relationship between pregnancy complications, such as preterm birth, miscarriage, or gestational conditions, and the onset of FHA will also be analyzed. Data will be collected through baseline and annual questionnaires throughout the study, providing a comprehensive understanding of these factors' roles in the development of FHA.

CONTACTS AND LOCATIONS:
Overall Officials: Chrisandra Shufelt, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No